CLINICAL TRIAL: NCT02294422
Title: Achieving Recommended Endotracheal Tube Cuff Pressure; A Randomized Control Trial Comparing Loss of Resistance Syringe to Pilot Balloon Palpation.
Brief Title: Balloon Palpation vs Loss of Resistance Syringe for Safe Endotracheal Tube Cuff Pressure; a Randomized Clinical Trial
Acronym: LOR-ETCP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Makerere University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2012/HD07/1766U
Record Dates: First submitted 2014-08-02; First posted 2014-11-19 (Estimated); Last update posted 2015-06-30 (Estimated); Status verified 2015-06

CONDITIONS: Tracheal Damage
Keywords: Loss of resistance; Pilot balloon; Cuff pressure; Endotracheal tube

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 2. LOR and aneroid manometer group (Experimental): after inflating the endotracheal tube (ETT) cuff using a loss of resistance syringe (BD Epillor LOR), the LOR syringe is left attached to the pilot balloon and and any excess pressure will be passively released until the plunger stops drawing back.
  Interventions: Device: LOR; Device: Aneroid manometer
- 1. PBP and aneroid manometer group (Placebo Comparator): The anaesthesia care provider shall inflate the ETT cuff via the pilot balloon with small volumes of air as he/she 'feels ' for the pressures in the pilot balloon to a pressure he/she thinks is just enough. An aneroid manometer (VBM, Germany. Accurate in the range 0-120 cmH2O +-2 cmH2O) shall then be attached by the investigator and measurement of the pressure taken.
  Interventions: Device: PBP; Device: Aneroid manometer

INTERVENTIONS:
Device: PBP — the pilot balloon is continuously palpated o felt for adequate pressure as its being inflated.
  Other Names: Pilot balloon palpation technique
  Arms: 1. PBP and aneroid manometer group
Device: LOR
  Other Names: LOR syinge
  Arms: 2. LOR and aneroid manometer group
Device: Aneroid manometer — The pilot balloon is attached onto the manometer and cuff pressures are raed off from the gauge.
  Other Names: VBM, Germany

SUMMARY:
This study is aimed at establishing whether use of loss of resistance syringe (LOR) that is traditionally used for identifying epidural space, is a better method for providing safe cuff pressures in adults intubated with cuffed endotracheal tubes. The conventional method is the use of pilot ballon palpation (PBP) to approximate cuff pressures but this is associated with airway damage.

The study hypothesis states that both the loss of resistance syringe method and the pilot balloon palpation methods achieve the recommended endotracheal tube intracuff pressures.

ELIGIBILITY:
Inclusion Criteria:

* American society of anesthesiologists (ASA) physical status classes I-IV

Exclusion Criteria:

* Known or anticipated laryngo-tracheal abnormalities.
* Patients with cough, sore throat, dysphagia and dysphonia.
* Patients in whom intubation is attempted more than twice

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Actual)
Dates: Start 2014-04; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
The percentage of subjects with intracuff pressure ranging from 20cm H2O to 30cmH2O | 5minutes
  This outcome will be measured within the first 5 minutes after intubation of the patient. The recommended range of intracuff pressure for this study is 20-30cmH2O

SECONDARY OUTCOMES:
Incidence of early postoperative airway symptoms | 12 hours
  Patents will be reviewed 12 hours after extubation for cough, sore throat, dysphagia and dysphonia.

CONTACTS AND LOCATIONS:
Overall Officials: Fred Bulamba, masters, Principal Investigator — Anaesthesiologist; Kintu Andrew, Fellowship, Study Chair — Lecturer; Arthur Kwizera, Masters, Study Director — Lecturer
Locations (1):
- Makerere University college of health sciences, Mulago National Referal Hospital Complex, Kampala, Uganda